CLINICAL TRIAL: NCT06352723
Title: Use of Cenobamate in the Intensive Care Unit for Acute Frequent Seizures and Status Epilepticus
Brief Title: Cenobamate in the Intensive Care Unit
Acronym: CENOBITE
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jong Woo Lee, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P000856
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Epilepsy; Neurologic Disorder
Keywords: ICU
MeSH Terms: conditions — Epilepsy; Nervous System Diseases | interventions — Cenobamate

STUDY DESIGN:
Intervention Model Description: Single arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cenobamate (Experimental): 400mg load plus 100mg a day for maximum of 14 days
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Study Drug: Cenobamate 400mg x 1 NGT/G-tube (Day 1), 100mg (Day 2-14)
  * Discontinued cenobamate upon cessation of seizures or RegiSCAR score 4-5 or at 14 days.
  * Adjust cenobamate dose based on patient response; this may include discontinuation if seizures resolve, or increase in dose to 150mg or 200mg a day after Day 7

SUMMARY:
The CENOBITE study will be conducted as a multi-center trial involving X leading centers from the Critical Care EEG Monitoring Consortium (CCEMRC). A total of 10 patients will be recruited over a period of one year, with each patient undergoing monitored treatment regimen. Each site will obtain its own approval from their institutional review board. Data will be shared through the MGB REDCap; raw EEG files will be shared through the MGB Dropbox and analyzed at the BWH.

Monitoring for the development of Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS) syndrome, a potential adverse reaction, will be a key aspect of the study. Regular assessments, including RegiSCAR scoring (a validated scoring system for DREeSS5), daily serum cenobamate level measurements, and comprehensive lab tests, will be conducted to ensure patient safety and the effective management of any adverse reactions such as DRESS syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70.
* Undergoing EEG monitoring.
* Acute frequent seizures (>1/hour) or status epilepticus (>5 min of consecutive seizures, or seizure burden >20% within past 1 hour).
* Adjunctive conventional antiseizure medication indicated.

Exclusion Criteria:

* History of medication-related rash.
* On medication or device affecting enteral absorption (e.g., phenobarbital, pentobarbital).
* Counterindication to cenobamate as described in the prescribing information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Target level | 6 hours after bolus
  Percentage of patients reaching target level of 10±2 ug/mL after load.
Maintenance level | Up to 14 days
  Percentage of patients maintaining daily therapeutic level of 10±2 ug/mL

SECONDARY OUTCOMES:
Seizure cessation | Up to 14 days
  Percentage of seizure cessation within 24 hours of reaching the target level.
Seizure burden change | Up to 14 days
  Percentage change in seizure burden over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Lee, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson JM, Molyneaux BJ, Lee JW. Safe Use of Cenobamate in Super Refractory Status Epilepticus: A Case Series. Neurohospitalist. 2023 Apr;13(2):169-172. doi: 10.1177/19418744221147083. Epub 2023 Feb 15. PMID 37064924